CLINICAL TRIAL: NCT02328742
Title: Pathophysiology of Intrauterine Synechia - Exploratory Study. Development of a Bioabsorbable Medical Device for the Prevention of Postoperative Intra-uterine Adhesions.
Brief Title: Development of a Bioabsorbable Medical Device for the Prevention of Postoperative Intra-uterine Adhesions.
Acronym: PréSynUT-1
Status: Withdrawn | Type: Observational
Why Stopped: Feasibility issues require solutions.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2013/VL-03; 2014-A00837-40 (Other: RCB number)
Record Dates: First submitted 2014-12-26; First posted 2014-12-31 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Infertility; Abortion, Spontaneous; Embryo Implantation, Delayed
MeSH Terms: conditions — Infertility; Abortion, Spontaneous | interventions — Hysteroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Endometrial biopsies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- No intracavitary pathology: During the first diagnostic hysteroscopy, patients in this group are found to not have an intracavitary pathology. (The first 20 such patients will be retained in this group.)
  Intervention: Hysteroscopy + endometrial biopsy
  Intervention: Telephone call
  Interventions: Biological: Hysteroscopy + endometrial biopsy; Other: Telephone call
- Synechia: During the first diagnostic hysteroscopy, patients in this group are found to have synechia.
  Intervention: Hysteroscopy + endometrial biopsy
  Intervention: Resection + endometrial biopsy
  Intervention: Follow-up hysteroscopy + endometrial biopsy
  Intervention: Telephone call
  Interventions: Biological: Hysteroscopy + endometrial biopsy; Other: Telephone call; Biological: Resection + endometrial biopsy; Biological: Follow-up hysteroscopy + endometrial biopsy
- Intracavitary pathology: During the first diagnostic hysteroscopy, patients in this group are found to have an intracavitary pathology.
  Intervention: Hysteroscopy + endometrial biopsy
  Intervention: Resection + endometrial biopsy
  Intervention: Follow-up hysteroscopy + endometrial biopsy
  Intervention: Telephone call
  Interventions: Biological: Hysteroscopy + endometrial biopsy; Other: Telephone call; Biological: Resection + endometrial biopsy; Biological: Follow-up hysteroscopy + endometrial biopsy

INTERVENTIONS:
Biological: Hysteroscopy + endometrial biopsy — The day of the first diagnostic hysteroscopy an endometrial biopsy is performed (biopsy A1). These biopsies will be used for the evaluation of TGFbeta, Activin A and inhibin.
  This intervention is required for the observational needs of this study.
Other: Telephone call — Patients will be contacted via telephone 6 months after first hysteroscopy.
  This intervention is required for the observational needs of this study.
Biological: Resection + endometrial biopsy — If patients are found to have synechia or another intracavitary pathology, resection is scheduled 1-2 months later. A second endometrial biopsy is performed at this time.
  This intervention is required for the observational needs of this study.
  Groups: Intracavitary pathology; Synechia
Biological: Follow-up hysteroscopy + endometrial biopsy — For patients having had resection, a follow-up hysteroscopy is performed 1 to 3 months later. An endometrial biopsy will be performed at this time.
  This intervention is required for the observational needs of this study.
  Groups: Intracavitary pathology; Synechia

SUMMARY:
The main objective of this study is to describe the level of expression of the biological factors involved in the formation of adhesions (Transforming growth factor beta, Activin A, inhibin) at the time of a first diagnostic hysteroscopy among women with synechia, another intracavitary disease or no intracavitary disease.

DETAILED DESCRIPTION:
The secondary obectives are:

A. For women who are found to have synechia or another intracavitary pathology at the time of resection: To describe the levels of Transforming growth factor beta, Activin A and Inhibin involved in synechia at the time of resection.

B. For women who are found to have synechia or another intracavitary pathology at the time of resection:To describe the levels of Transforming growth factor beta, Activin A and Inhibin involved in synechia at the time of a follow-up hysteroscopy following resection.

C. For women who are found to have synechia at the time of resection:To describe the change in levels of Transforming growth factor beta, Activin A and Inhibin involved at the time of a follow-up hysteroscopy following resection whether or not the patient converts back to "no synechia".

D. For women who are found to have another intracavitary pathology at the time of resection: To describe the change in levels of Transforming growth factor beta, Activin A and Inhibin involved at the time of a follow-up hysteroscopy following resection whether or not the patient converts to "synechia".

E. To estimate the intra-individual variation in the measured factors (initial biopsy levels versus levels at time of resection).

F. To create an intrauterine map of factor levels according to biopy position (riosteal / medium / proximal) for patients with synechia or another intracavitary pathology at the time of resection and then follow-up hysteroscopy.

G. To describe the levels of Transforming growth factor beta, Activin A and Inhibin as a function of pregnancy 6 months after resection.

H. Create a tissue bank associated with the study.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be given free and informed consent and must have signed the consent form
* The patient must be affiliated with or beneficiary of a health insurance plan
* Indication for hysteroscopy associated with one of the following: infertility evaluation, postoperative dysmenorrhea, embryo implantation failure after invitro fertilization, recurrent miscarriages

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, guardianship or curatorship
* The patient refuses to sign the consent
* It is not possible to correctly inform the patient
* The patient is postmenopausal
* Indication of hysteroscopy not associated with exploration of infertility or dysmenorrhea
* Presence of endometritis objectified via sampling during diagnostic hysteroscopy

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of women of childbearing age (≥18 years and <45 years) requiring a hysteroscopy motivated by an infertility evaluation, failure of embryo implantation after invitro fertilization, repeated miscarriages
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Activin A | Day 0 (day of diagnostic hysteroscopy)
Inhibin | Day 0 (day of diagnostic hysteroscopy)
Transforming growth factor beta | Day 0 (day of diagnostic hysteroscopy)
Diagnosis of synechia or other intracavitary pathology | Day 0 (day of diagnostic hysteroscopy)

SECONDARY OUTCOMES:
Activin A | 1 to 2 months after diagnostic hysteroscopy (day of resection)
Inhibin | 1 to 2 months after diagnostic hysteroscopy (day of resection)
Transforming growth factor beta | 1 to 2 months after diagnostic hysteroscopy (day of resection)
Diagnosis of synechia or other intracavitary pathology | 1 to 2 months after diagnostic hysteroscopy (day of resection)
Activin A | 1 to 3 months after resection (day of follow-up hysteroscopy)
Inhibin | 1 to 3 months after resection (day of follow-up hysteroscopy)
Transforming growth factor beta | 1 to 3 months after resection (day of follow-up hysteroscopy)
Diagnosis of synechia or other intracavitary pathology | 1 to 3 months after resection (day of follow-up hysteroscopy)
Pregnancy (yes/no) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Letouzey, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (3):
- France (3):
  - Institut des Biomolécules Max Mousseron, Montpellier
  - CHRU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes